CLINICAL TRIAL: NCT04798482
Title: Effect of Dexmedetomidine of Gastrointestinal Motility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Keira Mason, Associate Professor of Anaesthesia, Harvard Medical School Boston Children's Hospital, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00035865
Record Dates: First submitted 2021-02-18; First posted 2021-03-15 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dexmedetomidine (Experimental): This is a single arm, open label, interventional study examining the effects of dexmedetomidine on anal manometry. All subjects will be administered dexmedetomidine following their baseline manometry measurements. Following dexmedetomidine administration, anal manometry measurements will be observed for 15 minutes.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will undergo the usual anal manometry study, with no adjuvant medications, per routine practice currently in the gastrointestinal unit. Following completion of manometry, 0.5 mcg/kg DEX will be administered over 1 minute followed by an infusion of 0.15 mcg/kg/hr. Manometry measurements will be followed for 15 minutes in response to DEX.

SUMMARY:
Anorectal manometry requires that the patient be able to respond to command and not receive any medications which could alter muscle tone or motility. In the pediatric population, anorectal manometry can be psychologically challenging to parents and their child, as it is traditionally performed without adjuvant sedation or anesthesia. Sedatives and anesthesia can alter motility and smooth muscle activity, as well as render it difficult or impossible for the child to follow commands required of the study. Patient or parent non-compliance, inability to follow commands or to tolerate the procedure often renders the study invalid or impossible to complete. Dexmedetomidine is a sedative who's effect on anorectal musculature has not been studied nor determined. It would be important to determine whether it spares smooth muscle function, as it would provide a viable option to provide sedation to children while still preserving their ability to respond to command. The primary objective of this study is to examine the effects of dexmedetomidine on gastrointestinal smooth muscle by observing changes in anorectal manometry before and after dexmedetomdine administration.

DETAILED DESCRIPTION:
Primary objective:

To examine the effects of dexmedetomidine on intra-anal pressure and the dose response curve to balloon distention by comparing the baseline measurements with those after dexmedetomidine administration.

Dexmedetomidine is an alpha-2 agonist that is considered to be a smooth muscle relaxant. It's a potential use as a sedative for endoscopies has been considered. It is important to know whether or not it has effect on smooth muscle tone and would affect manometry studies in those patients who could receive it. The investigator hypothesizes that dexmedetomidine will have minimal effects in the dosing that is being administered.

Background:

Anorectal manometry requires that the patient be able to respond to command and not receive any medications which could alter muscle tone or motility. These patients typically have the manometry performed without any adjuvant sedatives, anesthetics or medications. In the pediatric population, anorectal manometry can be psychologically challenging to parents and their child, particularly without adjuvant sedation or anesthesia. There are some exceptional circumstances which require sedation/anesthesia administration for these procedures, either because the children are young (< 5 years), they have behavioral issues (like autism) or because they have severe anxiety. In those patients with severe issues even general anesthesia may be needed. The risk of administering any medication to these patients is that they can alter motility and smooth muscle activity, consequently artificially altering the results of the anal manometry. It is important to know which medications can be administered without affecting anal muscle tone. Dexmedetomidine is a newer sedative and anxiolytic. It could be valuable for anxiolysis for anal manometry. It's effect on anal smooth muscle, however, has never been studied. It would be important to determine whether it spares smooth muscle function, as it would provide a viable option to provide sedation to children while still preserving their ability to respond to command.

Dexmedetomidine is one of the standard drugs administered for sedation in children who require sedation for diagnostic (gastroendoscopic upper and lower procedures) and radiologic diagnostic imaging studies (MRI, CT and Nuclear Medicine). Over 17,000 infants, children and developmentally compromised young adults have been sedated with dexmedetomidine at Boston Children's Hospital without a cardiac or respiratory arrest, or a need to provide positive pressure assisted ventilation.

Methods:

Patients will undergo the usual anal manometry study, with no adjuvant medications, per routine practice currently in the gastrointestinal unit. Following completion of manometry, 0.5 mcg/kg DEX will be administered over 1 minute followed by an infusion of 0.15 mcg/kg/hr. Manometry measurements will be followed for 15 minutes in response to DEX.

Definition of Primary Endpoint:

Primary outcome: To examine the effects of dexmedetomidine on intra-anal pressure and the dose response curve to balloon distention by comparing the baseline measurements with those after dexmedetomidine administration. The pressure measurements will be recorded by the research team member who will be present, every 30 seconds starting from 5 minutes prior to DEX to 15 minutes following DEX administration.

Data Analysis Plan:

Data will be analyzed after the completion of the study. The manometry measurements will be done blindly by one of the investigators.

The following endpoints will be analyzed at the completion of the study: time to meet modified Aldrete discharge criteria, adverse events, need for unplanned airway interventions, intravenous anesthetic duration of sedation, presence of agitation/delirium (PAED score), and time of BIS score to return to baseline (pre-sedation level).

Statistical Power and Sample Considerations:

The study was powered and sample size calculated assuming a mean intra-anal pressure of 90 mmHg, with a mean reduction to 65 mmHg, and a standard deviation of 32. With a significance level of 0.05, it would require approximately 15 subjects to achieve power of 80.3%.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-18 years who are scheduled to have an anorectal manometry followed by an upper or lower endoscopic procedures at Boston Children's Hospital
* Patients are cooperative to do the anorectal manometry without sedation (besides pre-med midazolam)
* Anticipates to receive standard sedation with dexmedetomidine and propofol for a gastrointestinal procedure in the Gastroenterology Procedure Unit (GPU)
* Provides written consent to participate in the research study
* In females of reproductive age, pregnancy testing

Exclusion Criteria:

* Do not meet established sedation criteria
* Patients who require sedation prior to their anal manometry testing
* History of allergy, intolerance, or reaction to dexmedetomidine
* Current, repaired or risk of Moya-Moya disease
* Recent stroke (cerebrovascular accident) within past 6 months
* Uncontrolled hypertension
* Concomitant use of opioids, beta antagonist, alpha 2 agonist or calcium channel blocker
* BMI greater than 30 or weight above 110th percentile
* Refuses insertion of intravenous catheter while awake
* Currently receiving pharmacologic agents for hypertension or cardiac disease
* Currently receiving or has received digoxin within the past 3 months
* Active, uncontrolled gastroesophageal reflux (an aspiration risk), requiring endotracheal intubation.
* Current (or within past 3 months) history of apnea requiring an apnea monitor
* Unstable cardiac status (life threatening arrhythmias, abnormal cardiac anatomy, significant cardiac dysfunction)
* Craniofacial anomaly, which could make it difficult to effectively establish a mask airway for positive pressure ventilation if needed
* Active, current respiratory issues that are different from the baseline status (pneumonia, exacerbation of asthma, bronchiolitis, respiratory syncytial virus).

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keira Mason, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aantaa R, Kanto J, Scheinin M, Kallio A, Scheinin H. Dexmedetomidine, an alpha 2-adrenoceptor agonist, reduces anesthetic requirements for patients undergoing minor gynecologic surgery. Anesthesiology. 1990 Aug;73(2):230-5. doi: 10.1097/00000542-199008000-00007. PMID 1974394
- [Background] Ambartsumyan L, Rodriguez L, Morera C, Nurko S. Longitudinal and radial characteristics of intra-anal pressures in children using 3D high-definition anorectal manometry: new observations. Am J Gastroenterol. 2013 Dec;108(12):1918-28. doi: 10.1038/ajg.2013.361. Epub 2013 Oct 29. PMID 24169274
- [Background] Ozkose Z, Demir FS, Pampal K, Yardim S. Hemodynamic and anesthetic advantages of dexmedetomidine, an alpha 2-agonist, for surgery in prone position. Tohoku J Exp Med. 2006 Oct;210(2):153-60. doi: 10.1620/tjem.210.153. PMID 17023769
- [Background] Gurbet A, Basagan-Mogol E, Turker G, Ugun F, Kaya FN, Ozcan B. Intraoperative infusion of dexmedetomidine reduces perioperative analgesic requirements. Can J Anaesth. 2006 Jul;53(7):646-52. doi: 10.1007/BF03021622. PMID 16803911
- [Background] Pestieau SR, Quezado ZM, Johnson YJ, Anderson JL, Cheng YI, McCarter RJ, Choi S, Finkel JC. High-dose dexmedetomidine increases the opioid-free interval and decreases opioid requirement after tonsillectomy in children. Can J Anaesth. 2011 Jun;58(6):540-50. doi: 10.1007/s12630-011-9493-7. Epub 2011 Apr 2. PMID 21461792
- [Background] Le Guen M, Liu N, Tounou F, Auge M, Tuil O, Chazot T, Dardelle D, Laloe PA, Bonnet F, Sessler DI, Fischler M. Dexmedetomidine reduces propofol and remifentanil requirements during bispectral index-guided closed-loop anesthesia: a double-blind, placebo-controlled trial. Anesth Analg. 2014 May;118(5):946-55. doi: 10.1213/ANE.0000000000000185. PMID 24722260
- [Background] Morera C, Nurko S. Rectal manometry in patients with isolated sacral agenesis. J Pediatr Gastroenterol Nutr. 2003 Jul;37(1):47-52. doi: 10.1097/00005176-200307000-00008. PMID 12827005
- [Background] Sen S, Chakraborty J, Santra S, Mukherjee P, Das B. The effect of dexmedetomidine infusion on propofol requirement for maintenance of optimum depth of anaesthesia during elective spine surgery. Indian J Anaesth. 2013 Jul;57(4):358-63. doi: 10.4103/0019-5049.118558. PMID 24163449
- [Background] Al-Zaben KR, Qudaisat IY, Al-Ghanem SM, Massad IM, Al-Mustafa MM, Al-Oweidi AS, Abu-Halaweh SA, Abu-Ali HM, Saleem MM. Intraoperative administration of dexmedetomidine reduces the analgesic requirements for children undergoing hypospadius surgery. Eur J Anaesthesiol. 2010 Mar;27(3):247-52. doi: 10.1097/EJA.0b013e32833522bf. PMID 19952754
- [Background] Mason KP, Zurakowski D, Zgleszewski SE, Robson CD, Carrier M, Hickey PR, Dinardo JA. High dose dexmedetomidine as the sole sedative for pediatric MRI. Paediatr Anaesth. 2008 May;18(5):403-11. doi: 10.1111/j.1460-9592.2008.02468.x. Epub 2008 Mar 18. PMID 18363626
- [Background] Mason KP, Zgleszewski SE, Dearden JL, Dumont RS, Pirich MA, Stark CD, D'Angelo P, Macpherson S, Fontaine PJ, Connor L, Zurakowski D. Dexmedetomidine for pediatric sedation for computed tomography imaging studies. Anesth Analg. 2006 Jul;103(1):57-62, table of contents. doi: 10.1213/01.ane.0000216293.16613.15. PMID 16790626
- [Background] Heard C, Burrows F, Johnson K, Joshi P, Houck J, Lerman J. A comparison of dexmedetomidine-midazolam with propofol for maintenance of anesthesia in children undergoing magnetic resonance imaging. Anesth Analg. 2008 Dec;107(6):1832-9. doi: 10.1213/ane.0b013e31818874ee. PMID 19020127
- [Background] Kol IO, Egilmez H, Kaygusuz K, Gursoy S, Mimaroglu C. Open-label, prospective, randomized comparison of propofol and sevoflurane for laryngeal mask anesthesia for magnetic resonance imaging in pediatric patients. Clin Ther. 2008 Jan;30(1):175-81. doi: 10.1016/j.clinthera.2008.01.008. PMID 18343254
- [Background] Koroglu A, Teksan H, Sagir O, Yucel A, Toprak HI, Ersoy OM. A comparison of the sedative, hemodynamic, and respiratory effects of dexmedetomidine and propofol in children undergoing magnetic resonance imaging. Anesth Analg. 2006 Jul;103(1):63-7, table of contents. doi: 10.1213/01.ANE.0000219592.82598.AA. PMID 16790627
- [Background] Cravero JP, Beach ML, Blike GT, Gallagher SM, Hertzog JH; Pediatric Sedation Research Consortium. The incidence and nature of adverse events during pediatric sedation/anesthesia with propofol for procedures outside the operating room: a report from the Pediatric Sedation Research Consortium. Anesth Analg. 2009 Mar;108(3):795-804. doi: 10.1213/ane.0b013e31818fc334. PMID 19224786
- [Background] Bassett KE, Anderson JL, Pribble CG, Guenther E. Propofol for procedural sedation in children in the emergency department. Ann Emerg Med. 2003 Dec;42(6):773-82. doi: 10.1016/s0196-0644(03)00619-x. PMID 14634602
- [Background] Guenther E, Pribble CG, Junkins EP Jr, Kadish HA, Bassett KE, Nelson DS. Propofol sedation by emergency physicians for elective pediatric outpatient procedures. Ann Emerg Med. 2003 Dec;42(6):783-91. doi: 10.1016/s0196-0644(03)00634-6. PMID 14634603
- [Background] Hauber JA, Davis PJ, Bendel LP, Martyn SV, McCarthy DL, Evans MC, Cladis FP, Cunningham S, Lang RS, Campbell NF, Tuchman JB, Young MC. Dexmedetomidine as a Rapid Bolus for Treatment and Prophylactic Prevention of Emergence Agitation in Anesthetized Children. Anesth Analg. 2015 Nov;121(5):1308-15. doi: 10.1213/ANE.0000000000000931. PMID 26332857
- [Background] Nafiu OO, Kheterpal S, Morris M, Reynolds PI, Malviya S, Tremper KK. Incidence and risk factors for preincision hypotension in a noncardiac pediatric surgical population. Paediatr Anaesth. 2009 Mar;19(3):232-9. doi: 10.1111/j.1460-9592.2008.02871.x. Epub 2008 Dec 1. PMID 19143955
- [Background] Anderson JL, Junkins E, Pribble C, Guenther E. Capnography and depth of sedation during propofol sedation in children. Ann Emerg Med. 2007 Jan;49(1):9-13. doi: 10.1016/j.annemergmed.2006.06.011. Epub 2006 Aug 17. PMID 17141136
- [Background] Miller P, Mack CD, Sammer M, Rozet I, Lee LA, Muangman S, Wang M, Hollingworth W, Lam AM, Vavilala MS. The incidence and risk factors for hypotension during emergent decompressive craniotomy in children with traumatic brain injury. Anesth Analg. 2006 Oct;103(4):869-75. doi: 10.1213/01.ane.0000237327.12205.dc. PMID 17000796
- [Background] Chandran V, Jagadisan B, Ganth B. Validation of Adapted Dartmouth Operative Conditions Scale for sedation during pediatric esophagogastroduodenoscopy. Paediatr Anaesth. 2017 Jun;27(6):621-628. doi: 10.1111/pan.13127. Epub 2017 Apr 3. PMID 28370856

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexmedetomidine
Started | 22
Completed | 20
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Lost eligibility | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.29 (4.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: American | 13
  Ethnicity: French | 1
  Ethnicity: Arabic | 1
  Ethnicity: Canadian | 1
  Ethnicity: English | 1
  Ethnicity: Unknown | 5
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Intra-anal Sphincter Pressure (IASP) 1 Minute After Dexmedetomidine Administration
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 20
mmHg | 62.9 (4.5)

2. Primary Outcome: Intra-anal Sphincter Pressure (IASP) 5 Minutes After Dexmedetomidine Administration
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 20
mmHg | 45.1 (3.7)

3. Primary Outcome: Intra-anal Sphincter Pressure (IASP) Baseline Measurement
Description: IASP recorded prior to administration of dexmedetomidine
Time Frame: 30 seconds
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dexmedetomidine
Number analyzed (Participants) | 20
mmHg | 80.5 (5.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on the day of the procedure, during study involvement and immediately following in the post-anesthesia care unit. Subjects were monitored for AEs for 1 day.
Arm/Group | Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT04798482/Prot_SAP_000.pdf